CLINICAL TRIAL: NCT02204358
Title: Clinical Study of the Treatment of Infertility Caused by Severe Intrauterine Adhesions by Collagen Scaffold Loaded With Autologous Bone Marrow Stem Cells
Brief Title: Treatment of Infertility by Collagen Scaffold Loaded With Autologous Bone Marrow Stem Cells
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yali Hu, MD,PhD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012022
Record Dates: First submitted 2014-07-26; First posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Infertility; Intrauterine Adhesions; Endometrial Dysplasia
MeSH Terms: conditions — Infertility; Gynatresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous bone marrow stem cells (Experimental): Using collagen scaffold loaded with autologous bone marrow stem cells to treat severe intrauterine adhesions or endometrial dysplasia.
  Interventions: Procedure: autologous bone marrow stem cells

INTERVENTIONS:
Procedure: autologous bone marrow stem cells — Before considering whether patients meet the inclusion criteria, they are diagnosed with severe intrauterine adhesions uterus, endometrial dysplasia. And after that there will be history taking, physical examination, chromosome examination, B-ultrasound examination, hysteroscopy examination and so on.
  If patients agree to participate, they will receive a bone marrow stem cells collection and separation of adhesions by hysteroscopy surgery. Postoperative observation period is about three months, including B-ultrasound examination once a month and hysteroscopy after 3 months. According to the endometrial conditions, the doctor will select an appropriate time for pregnancy and follow-up. The doctor may also require patients to do some unscheduled visits.
  Other Names: infertility; severe intrauterine adhesions; endometrial dysplasia; collagen scaffold

SUMMARY:
Study of the treatment of infertility caused by severe intrauterine adhesions or endometrial dysplasia by collagen scaffold loaded with autologous bone marrow stem cells, and to provide clinical evidence for the treatment of uterine infertility

DETAILED DESCRIPTION:
Infertility is defined as a women fails to become pregnant after having a normal sex life for two years without contraception. There is no effective treatment to the infertility caused by severe intrauterine adhesions or endometrial dysplasia which affects embryos implantation. The existing drugs, physical or surgical treatments had no significant effects to severe intrauterine adhesions.Collagen is the main component of the extracellular matrix with good biocompatibility, and it has been approved for the reparation of skin and oral mucosa by State Food and Drug Administration. Bone marrow stem cells have been used in the clinical treatment of blood diseases, and achieved good results. In this study, collagen scaffold and autologous bone marrow stem cells are combined, and they showed good biological safety

ELIGIBILITY:
Inclusion Criteria:

* Infertility caused by serious intrauterine adhesions or endometrial dysplasia
* Hysteroscopy examination confirmed intrauterine adhesions or endometrial dysplasia
* Monitoring of endometrial cycle
* Sign a consent form
* Follow the test plan and follow-up process

Exclusion Criteria:

* Abnormal chromosome karyotype
* Congenital uterine malformations
* Severe endometriosis
* Severe adenomyosis
* Contraindications to pregnancy
* Contraindications to bone marrow collection
* Contraindications to hormone replacement therapy
* Medical history of pelvic tumors or receiving pelvic radiotherapy
* Unable to adhere to the hospital examination and follow-up, or carrying on other treatment during follow-up period

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of intrauterine scar area,the change of intrauterine adhesion | up to 3 months
  hysteroscope ,understanding improvement of uterine cavity form,the degree and nature of adhesion or the vanishment of intrauterine adhesion,and the reduction of scar and its area,comparing with pre-operation

SECONDARY OUTCOMES:
The change of endometrial thickness | up to 1 month
  Measure the endometrial thickness and endometrial blood supply during ovulation by ultrasound by the same trained medical sonographers,comparing with pre-operation.
The change of endometrial thickness | up to 2 months
  Measure the endometrial thickness and endometrial blood supply during ovulation by ultrasound by the same trained medical sonographers,comparing with pre-operation.
menstrual blood volume The change of menstrual blood volume | baseline and 1 month
  Understanding the menstrual blood volume after surgery ,the number of sanitary napkins per day ,and number of days,comparing with pre-operation.

OTHER OUTCOMES:
rate of pregnancy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yali HU, MD,PhD, Principal Investigator — Vice-president of the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China